CLINICAL TRIAL: NCT05185739
Title: PRIMER-1 Perioperative Pembrolizumab and Lenvatinib in Resectable Hepatocellular Carcinoma (HCC)
Brief Title: Perioperative Pembrolizumab and Lenvatinib in Resectable Hepatocellular Carcinoma (HCC)
Acronym: PRIMER-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/12/6928
Record Dates: First submitted 2021-11-02; First posted 2022-01-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver cancer,; pembrolizumab; lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: This is a randomised 3-arm phase II clinical trial in patients with resectable HCC. Sixty patients will be randomized 1:1:1 to pembrolizumab, lenvatinib or the combination of pembrolizumab and lenvatinib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab (Active Comparator)
  Interventions: Drug: Pembrolizumab
- Lenvatinib. (Active Comparator)
  Interventions: Drug: Lenvatinib
- Pembrolizumab and Lenvatinib. (Experimental)
  Interventions: Drug: Pembrolizumab and Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Pre-operative Pembrolizumab (200mg IV every 3 weeks) for 2 cycles
  Arms: Pembrolizumab
Drug: Lenvatinib — Pre-operative Lenvatinib (8 or 12mg PO once daily according to bodyweight <60gk≥) for 6 weeks
  Arms: Lenvatinib.
Drug: Pembrolizumab and Lenvatinib — Pre-operative combination of pembrolizumab and lenvatinib at the standard doses and duration as per cohort 1 and 2
  Arms: Pembrolizumab and Lenvatinib.

SUMMARY:
This is a multicentre randomised 3-arm phase II clinical trial in patients with resectable Hepatocellular Carcinoma (HCC). Sixty patients will be randomized 1:1:1 to 6 weeks of pre-operative therapy with: pembrolizumab, lenvatinib or the combination of pembrolizumab and lenvatinib followed by up to 12 months treatment with post-operative pembrolizumab. The aim of the study is to compare the efficacy of pembrolizumab combined with lenvatinib with that of pembrolizumab and lenvatinib alone in terms of major pathological response in patients with resectable HCC. Major pathological response will be defined by the proportion of patients with less than 10% viable tumour at resection.

DETAILED DESCRIPTION:
Hepatocellular Carcinoma (HCC), or Liver cancer, is the second most common cause of cancer-related death worldwide and is the most rapidly increasing cause of cancer-related death in the West. The only potentially curative options are transplantation, surgical resection and ablation. Both surgical resection and ablation are associated with a high rate of recurrence and 70% of resected patients relapse within 5 years. To date, no standard adjuvant therapies have been approved. Recent studies provide evidence that immunotherapy may address a significant unmet need in the management of HCC.

Furthermore, there is also a rationale for pre-operative therapy which has been shown to be superior to a postoperative treatment approach as supported by pre-clinical studies. The feasibility and outcomes of this approach have recently been reported in the setting of lung cancer. Lenvatinib, an immunotherapy drug, has been approved as a first treatment option in HCC. Pembrolizumab, another immunotherapy treatment has been evaluated as first treatment option in HCC in two clinical trials. The combination of these two drugs has been explored in HCC in early phase trials.

The aim is to compare the efficacy of pembrolizumab (a type of immunotherapy designed to 're-awaken' the immune system) combined with lenvatinib (an anti-cancer drug that is a multiple kinase inhibitor) with that of pembrolizumab and lenvatinib alone in patients with resectable Hepatocellular Carcinoma.

Treatment lasts for up to 18 months. Depending on when patients are recruited, patients will be followed up for a minimum of 1 year and maximum of 3 years, following the end of their post-surgery treatment. It is expected that it will take 24 months to recruit all the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of Hepatocellular Carcinoma (HCC) confirmed by radiology, histology, or cytology (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible) and suitable for surgical resection. Radiological confirmation of diagnosis is provided by the study site and defined by the presence of a liver mass of at least 1 cm and exhibiting arterial hypervascularity with washout in the portal venous phase seen in a tri-phasic magnetic resonance imaging (MRI).
2. Measurable disease based on RECIST 1.1
3. HCC amenable to R0 resection with curable intent
4. Child-Pugh A liver disease
5. International normalised ratio (INR) ≤1.4
6. ECOG Performance status 0 or 1
7. Adequate haematological function as defined by:

   * Haemoglobin (Hb) > 90g/l
   * Neutrophil Count > 1.5 x 109/l
   * Platelets > 75 x 109/l
8. Adequate renal function with GFR >40ml/min using a validated creatinine clearance calculation (e.g. Cockcroft-Gault or Wright formula)
9. Adequate liver function as defined by:

   * Aminotransferase (ALT) or aspartate aminotransferase (AST) < 5.0 x ULN
   * Albumin >32g/l
   * Amylase ≤ 1.5 x ULN
10. Patients with past or ongoing hepatitis C virus (HCV) infection will be eligible for the study if HCV viral load is undetectable at screening. The treated patients must have completed their treatment curative anti-viral treatment at least 4 weeks prior to randomisation.
11. Patients with controlled hepatitis B will be eligible as long as they meet the following criteria:

    * Antiviral therapy for hepatitis B virus (HBV) must be given for at least 4 weeks and HBV viral load must be less than 500 IU/mL prior to randomisation. Patients on active HBV therapy with viral loads under 500 IU/mL should stay on the same therapy throughout study treatment.
    * Patients who are positive for anti-hepatitis B core antibody (HBc), negative for hepatitis B surface antigen (HBsAg), and negative or positive for anti-hepatitis B surface antibody (HBs), and who have an HBV viral load under 500 IU/mL, do not require HBV anti-viral prophylaxis
12. 18 years of age or over
13. Predicted life expectancy of > 3 months
14. Patients must have given written informed consent
15. Patients must have the ability to swallow oral medication
16. Must be willing to use effective contraception during study for 120 days after last dose.

Exclusion Criteria:

1. Has received any systemic chemotherapy, including anti-VEGF therapy, or any systemic investigational anticancer agents for advanced/unresectable HCC.
2. Has received local therapy including trans arterial embolic, chemo- or radiotherapy, external beam radiotherapy or ablative therapy to the measurable lesion to be resected.
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, or CD137).
4. Oesophageal or gastric variceal bleeding within the last 6 months.
5. Has received a live vaccine within 30 days prior to registration (seasonal flu vaccines that do not contain live virus are permitted). Administration of killed vaccines is allowed.
6. Active autoimmune disease that has required systemic treatment (i.e., with use of disease-modifying agents, corticosteroids or immunosuppressive drugs) in past 2 years except

   * Vitiligo
   * Psoriasis
   * Autoimmune-related hyperthyroidism
   * Autoimmune-related hypothyroidism who are in remission or on a stable dose of thyroid-replacement hormone replacement therapy (e.g., levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
7. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
8. A diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10mg daily prednisolone equivalent) or any other form of immunosuppressive therapy within 7 days prior to treatment.
9. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
10. Has clinical or radiological evidence of ascites on physical examination that is not controlled with medication.
11. Uncontrolled blood pressure (Systolic BP)>150 mmHg or diastolic BP >90 mmHg) with no change in anti-hypertensive medications within 1 week prior to randomisation.
12. Has had clinically diagnosed hepatic encephalopathy in the last 6 months.
13. Has medical contraindications that preclude all forms of contrast enhanced imaging (tri-phasic CT or MRI).
14. Gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
15. Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
16. Clinically significant haemoptysis from any source or tumour bleeding within 2 weeks prior to start of treatment.
17. Electrolyte abnormalities that have not been corrected.
18. Significant cardiovascular impairment within 12 months of start of treatment such as history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of start of treatment, or cardiac arrhythmia requiring medical treatment at screening.
19. Prolongation of QTc interval to > 480 ms.
20. Left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO).
21. Patients who are at risk for severe haemorrhage, bleeding or thrombotic disorders, or are receiving factor X inhibitors or anticoagulants that require therapeutic INR monitoring e.g. warfarin or similar agents. The degree of tumour invasion/infiltration of major blood vessels should be considered because of the potential risk of severe haemorrhage associated with tumour shrinkage/necrosis following lenvatinib therapy.
22. Patients having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
23. Patients who have not recovered adequately from any toxicity from other anti- cancer treatment regimens and/or complications from major surgery prior to starting therapy.
24. Has had major surgery to the liver prior to start of treatment. Note: If patient received any major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
25. Has had a minor surgery (i.e., simple excision) within 7 days prior to start of treatment (Cycle 1 Day 1).
26. Has a serious non-healing wound, ulcer, or bone fracture.
27. History of human immunodeficiency virus (HIV) infection.
28. Has an active infection requiring systemic therapy, with the exception of HBV, HCV.
29. Has severe hypersensitivity (≥Grade 3) to pembrolizumab or lenvatinib and/or any of their excipients.
30. Has dual active HBV infection (HBsAg (+) and /or detectable HBV DNA) and HCV infection (anti-HCV Ab (+) and detectable HCV RNA) at study entry.
31. Has dual active HBV infection and hepatitis D virus (HDV) at the study entry.
32. Has a known history of active tuberculosis (Bacillus tuberculosis).
33. Has a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the study.
34. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention. Note: Patients who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
35. Has had an allogenic tissue/solid organ transplant.
36. Women who are pregnant or breast feeding.
37. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
38. Have extra-hepatic spread or macrovascular invasion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate, defined as the proportion of patients with less than 10% viable tumour at resection. | At 4 months
  The primary aim of the study is to test the hypothesis that the combination of pembrolizumab and lenvatinib result in a higher rate of major pathological response than either drug used as a single-agent in patients with resectable hepatocellular carcinoma.

SECONDARY OUTCOMES:
Percentage of viable tumour cells at resection | At 4 months
  The primary aim of the study is to test the hypothesis that the combination of pembrolizumab and lenvatinib result in a higher rate of major pathological response than either drug used as a single-agent in patients with resectable hepatocellular carcinoma.
Radiological response rate | Evaluated pre-surgery (at 2 months)
  The hypothesis is that the radiological response rate of pembrolizumab and lenvatinib in combination is greater than that of pembrolizumab and lenvatinib as single agents. Measured by RECIST 1.1 and mRECIST performed pre-operatively and compared with pre-treatment baseline imaging)
Relapse free survival at 12 months from surgery | 12 months from surgery
  Relapse free survival at 12 months from surgery
Proportion of patients with surgery delayed by more than 4 weeks from the planned surgery date | Evaluated by time to surgery (at 3 months)
  Defined as the proportion of patients with surgery delayed by more than 4 weeks from the planned surgery date due to IMP-related adverse events (AEs) or serious adverse events (SAEs))
30-day post-operative surgical complication rate | Evaluated 30 days post surgery
  based on the Clavien-Dindo classification
Completion of protocol-defined therapy | 6 weeks pre-operative
  measured by the proprtion of patients mpleting protocol defined study-drug intervention.
Completion of protocol-defined therapy | 12 months post-operative
  measured by the proprtion of patients mpleting protocol defined study-drug intervention.
Determine the toxicity of pre-operative therapy according to Common Terminology Criteria for Adverse Events (CTCAE) V5. | Evaluated by monthly follow-up until patient relapse/ maximum of 3 years, following the end of their post-surgery treatment.
  Incidence and of adverse events (AEs) reported. Events will be classified according to CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tim Meyer, BSc MBBS PhD FRCP, Principal Investigator — University College, London
Locations (11):
- United Kingdom (11):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's Hospital, Leeds
  - Clatterbridge Cancer Centre, Liverpool
  - Hammersmith Hospital, London
  - King's College Hospital, London
  - Royal Free Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne